CLINICAL TRIAL: NCT05505838
Title: Expanded Access Protocol to Provide Patisiran to Patients With Transthyretin-mediated Amyloidosis (ATTR Amyloidosis) With Cardiomyopathy
Brief Title: Expanded Access Protocol to Provide Patisiran to Patients With Transthyretin-mediated Amyloidosis With Cardiomyopathy
Status: No longer available | Type: Expanded Access
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTR02-014
Record Dates: First submitted 2022-08-11; First posted 2022-08-18 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Transthyretin-mediated Amyloidosis With Cardiomyopathy; ATTR Amyloidosis With Cardiomyopathy
Keywords: RNAi therapeutic; Amyloidosis; Cardiomyopathy; TTR; Transthyretin
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies | interventions — patisiran

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Patisiran — Patisiran administered by intravenous (IV) infusion
  Other Names: ONPATTRO; ALN-TTR02

SUMMARY:
The objective of the study is to assess the long-term safety of patisiran in patients with ATTR amyloidosis with cardiomyopathy as assessed by a review of adverse events (AEs).

DETAILED DESCRIPTION:
Choosing to participate in an expanded access program is an important personal decision. Talk with your doctor and family members or friends about deciding to join a research study. To learn more about this study, please have your doctor contact the study research staff using the Contacts provided.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of ATTR amyloidosis with cardiomyopathy, classified as either hATTR amyloidosis with cardiomyopathy or wtATTR amyloidosis with cardiomyopathy; AND

  * Had an inadequate response to or could not tolerate standard of care, in the opinion of the investigator.
* Is not eligible for on-label use of commercial patisiran in the opinion of the investigator.

Exclusion Criteria:

* New York Heart Association (NYHA) Class IV
* NYHA Class III AND ATTR amyloidosis disease Stage 3 (defined as both N-terminal prohormone B-type natriuretic peptide (NT-proBNP) >3000 ng/L and estimated glomerular filtration rate [eGFR] <45 ml/min/1.73 m^2). [Gillmore 2018]
* Current or future participation in another investigational device or drug study, scheduled to occur during this study, or has received an investigational agent or device within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to dosing (Day 1). Patients who have previously participated in a gene therapy trial for hATTR amyloidosis.
* Patients currently enrolled in, eligible for inclusion in, or who have dropped out of an ongoing interventional (therapeutic) clinical trial related to ATTR amyloidosis.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (20):
- United States (20):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - NorthShore University, Evanston, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Penn Presbyerian Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - University of Utah, Salt Lake City, Utah